CLINICAL TRIAL: NCT06340711
Title: Phase II Study of Suratadenoturev (OBP-301) in Combination With Pembrolizumab in Immunotherapy Refractory Esophagogastric Adenocarcinoma
Brief Title: Study of Suratadenoturev (OBP-301) in Combination With Pembrolizumab in Esophagogastric Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Oncolys BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-06026219
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Adenocarcinoma; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Pembrolizumab; OBP-301; Immunotherapy
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OBP-301 Plus Pembrolizumab (Experimental): All participants will receive 4 intratumoral injections of OBP-301 with each injection occurring approximately 2 weeks apart. All participants will also receive infusions of pembrolizumab every 6 weeks until disease progression or for a maximum of 2 years.
  Interventions: Drug: OBP-301; Drug: Pembrolizumab

INTERVENTIONS:
Drug: OBP-301 — 2×10(12) viral particles per injection given intratumorally every 2 weeks for a total of 4 injections starting on Day 1 of the study
  Other Names: Suratadenoturev
Drug: Pembrolizumab — 400 mg IV given every 6 weeks starting on day 4 of the study and given for up to 2 years
  Other Names: Keytruda

SUMMARY:
The goal of this study is to learn about of the research study drug, telomelysin (OBP-301), in combination with pembrolizumab in advanced or metastatic gastric or gastroesophageal junction (GEJ) cancer. The main question it aims to answer is whether this combination is safe and effective in this type of cancer.

Participants will receive 5 injections of OBP-301, approximately every 2 weeks. OBP-301 will be injected directly into the tumor during an esophagogastroduodenoscopy (EGD). At the same time as the injection, a tumor biopsy will be taken. Participants will also receive pembrolizumab infusions every 6 weeks until disease progression or for a maximum of two years. Pembrolizumab infusions will occur on different days than OBP-301 injections.

DETAILED DESCRIPTION:
This is a phase II study of suratadenoturev (OBP-301) with pembrolizumab in advanced or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma that has progressed on at least 1 line of prior therapy for advanced disease. Patients must have received prior immunotherapy (anti PD-1 therapy). This study will examine the addition of OBP-301 with pembrolizumab patients who are refractory to first line immunotherapy.

Patients will undergo intra-tumoral injection of OBP-301 followed 2-4 days later by the administration of pembrolizumab. The OBP-301 injection will then be repeated every two weeks for 4 planned treatments, and up to one additional optional treatment. Pembrolizumab will be administered every 6 weeks until disease progression.

The primary endpoint is objective response rate, with the target response rate of 20%, to examine the hypothesis that OBP-301 can overcome checkpoint resistance. The expected response to continuing anti-PD-1 therapy in this patient population would anticipated to be <5%. As a key secondary endpoint, the investigators will also examine duration of response and progression free survival. In a previous trial of OBP-301 and pembrolizumab in the third line setting, two patients who had a partial response are now off therapy and without evidence of disease, with a duration of response 33+ months and 20+ months. The third patient with a partial response has been on therapy for 15+ months.

This trial utilizes a Simon's two-stage Minimax design. In the first stage of the trial, 13 patients will be accrued. If there are 0 responses in these 13 patients, the study will be stopped. Otherwise, 14 additional patients will be accrued for a total of 27 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma amenable to intra-tumoral injection (i.e. at least 1 cm in size)
* Tumor must be PD-L1 positive as defined by a combined positive score (CPS), i.e. CPS ≥ 1 by approved, commercial diagnostic assay
* Tumor must be HER2 negative as determined by a CLIA-approved laboratory

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 3 weeks of study Day 1.
* Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (greater than equivalent of 20 mg/day) or any other form of immunosuppressive therapy within 7 days prior to study Day 1.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has had prior anti-cancer monoclonal antibody chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1, who has not recovered from adverse events due to a previously administered agent.
* Has a known additional malignancy within 3 years before the first OBP-301 administration that is progressing or requires active treatment, with the exception of prostate cancer controlled with androgen deprivation therapy.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Is known to have acute or chronic active hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy within 2 weeks of Day 1.
* Is unable to comply with protocol procedures
* Previous severe hypersensitivity (≥ Grade 3) to any monoclonal antibody
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has had an allogenic tissue/solid organ transplant
* Has certain uncontrolled illnesses
* Is pregnant or breastfeeding or planning to become pregnant or start breast feeding during the study time period
* Is expecting to get someone else pregnant during the study time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Overall response rate as assessed by the RECIST v1.1 | Until disease progression or death, or for a maximum of approximately 2 years
  Overall response is defined as the sum of partial responses plus complete responses as defined by RECIST v1.1 criteria.
Number of serious adverse events (SAEs) tabulated by severity and classification per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 | Until 90 days after the last dose of study drug
  All SAEs will be recorded and coded by CTCAE v5 term and reported by severity and potential relatedness to study drugs
Number of adverse events (AEs) tabulated by severity and classification per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 | Until 30 days after the last dose of study drug
  All AEs will be recorded and coded by CTCAE v5 term and reported by severity and potential relatedness to study drugs

SECONDARY OUTCOMES:
Disease control rate (DCR) | Until disease progression or death, for a maximum of approximately 2 years from start of treatment
  Disease control rate is defined as the percentage of patients who have achieved complete response, partial response or stable disease.
Duration of response (DoR) | Until disease progression or death, or for a maximum of approximately 2 years from start of treatment
  Duration of response is defined as the duration that subjects who have responded to combination therapy remain without disease progression
Overall Survival (OS) | Until death or a maximum of 96 weeks from end of treatment (for a maximum of approximately 4 years from start of treatment)
  Overall Survival is defined as the time from registration to death due to any cause.
Progression free survival (PFS) | Until disease progression or death, or for a maximum of approximately 2 years from start of treatment
  Progression-free survival (PFS) is defined as time from registration to progression or death due to any cause. Progression is defined as radiologic progression of disease by RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No